CLINICAL TRIAL: NCT06733597
Title: Femoral Bone Mineral Density (BMD) Change Following Cemented or Cementless Total Knee Arthroplasty
Brief Title: Femoral BMD Change Following Cemented or Cementless Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-0197; Protocol Version 1/9/2026 (Other: UW Madison); A536110 (Other: UW Madison)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthropathy
Keywords: bone mineral density
MeSH Terms: interventions — Dental Cements; Robotic Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cemented and Manual (Active Comparator)
  Interventions: Procedure: Cement; Procedure: Manual Surgery
- Cemented and Robotic (Active Comparator)
  Interventions: Procedure: Cement; Procedure: Robotic Surgery
- Cementless and Manual (Active Comparator)
  Interventions: Other: Cementless; Procedure: Manual Surgery
- Cementless and Robotic (Active Comparator)
  Interventions: Other: Cementless; Procedure: Robotic Surgery

INTERVENTIONS:
Procedure: Cement — The cemented approach includes inserting cement into the femur and tibia prior to setting the prosthetic.
  Arms: Cemented and Manual; Cemented and Robotic
Other: Cementless — The non-cement approach uses a different type of prosthetic that is placed tight against the bone and requires no other fixation material.
  Arms: Cementless and Manual; Cementless and Robotic
Procedure: Manual Surgery — The manual approach is the surgeon determining prosthetic placement using techniques developed during training.
  Arms: Cemented and Manual; Cementless and Manual
Procedure: Robotic Surgery — The haptic robotic assisted approach uses a computer and robot to determine specific placement of the prosthetic.
  Arms: Cemented and Robotic; Cementless and Robotic

SUMMARY:
The purpose of this study is to examine femur bone mineral density (BMD) change before and after surgery in patients receiving cemented or cementless total knee arthroplasty (TKA). performed with manual or robotic methods. 100 participants will be enrolled and can expect to be on study for up to 26 months.

DETAILED DESCRIPTION:
It has previously been reported that total knee arthroplasty (TKA) causes major femur bone loss (~18% within 1 year). Prior studies did not examine different surgical methods, such as the use of cement or robotics, in TKA. The investigators hypothesize that previously reported differences in distal femur BMD change following TKA exist between patients receiving cemented vs. cementless prostheses.

Specific Aim 1: In the entire study cohort, our primary endpoint is to estimate percent BMD change 12 and 24 months after TKA at the distal femur 25% region of interest (ROI).

Specific Aim 1a: To compare percent BMD change 12 and 24 months after TKA at the distal femur 25% ROI in cemented vs uncemented implants.

Specific Aim 1b: To compare percent BMD change 12 and 24 months after TKA at the distal femur 25% ROI in those receiving robotic vs manual implants.

Specific Aim 2: In the entire study cohort, our secondary endpoints are to estimate percent BMD change 12 and 24 months after TKA at a.) the distal femur 15% ROI and b.) a proximal tibial ROI Specific Aim 2a: To compare percent BMD change 12 and 24 months after TKA at the distal femur 15% ROI and proximal tibial ROI in cemented vs uncemented implants.

Specific Aim 2b: To compare percent BMD change 12 and 24 months after TKA at the distal femur 15% ROI and proximal tibial ROI in in those receiving robotic vs manual implants.

Exploratory Aim 1: Compare patient reported pain and function at 2 weeks, 3 months, 12 months, and 24 months;

1. in those receiving cemented and cementless implants.
2. in those receiving robotic vs manual implants.

Exploratory Aim 2: Evaluate leg lean mass change as measured by DXA and BIS at 2 weeks, 3 months, 12 months, and 24 months over time.

1. In the entire cohort
2. in those receiving cemented and cementless implants.
3. in those receiving robotic vs manual implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than or equal to 55 years undergoing TKA with no prior total joint arthroplasty on the surgical side
* Normal BMD or osteopenia with Fracture Risk Assessment Tool (FRAX) not meeting Bone Health and Osteoporosis Foundation (BHOF) treatment recommendations, i.e., 10-year major osteoporotic fracture risk greater then or equal to 20 percent or hip fracture risk greater than or equal to 3 percent.

Exclusion Criteria:

* Known clinical osteoporosis defined as any one of the following:

  * Hip or spine T-score less than or equal to -2.5
  * History of low trauma fracture after age 50
  * FRAX fracture risk calculation greater than or equal to 20 percent for major osteoporotic fracture or greater than or equal to 3 percent for hip fracture
* Prior or current use of osteoporosis medications
* Current use of systemic glucocorticoids or bone-active medications
* Rheumatoid arthritis
* Laboratory abnormalities that in the opinion of study investigators may impact bone mineral density; including calcium, creatinine, albumin and parathyroid hormone (PTH)
* 25(OH)D less than 20 ng/mL
* Not suitable for study participation due to other reasons at the investigator's discretion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density within 25 percent of the region of interest at 12 and 24 months post TKA: All Participants | 12 months, 24 months
  Primary endpoint is to estimate percent BMD change 12 and 24 months after TKA at the distal femur, 25 percent region of interest, reported for all participants together.
Percent Change in Bone Mineral Density within 25 percent of the region of interest at 12 and 24 months post TKA: Cemented vs Uncemented | 12 months, 24 months
  Compare percent BMD change 12 and 24 months after TKA at the distal femur, 25 percent region of interest between all cemented and uncemented implants.
Percent Change in Bone Mineral Density within 25 percent of the region of interest at 12 and 24 months post TKA: Robotic vs Manual | 12 months, 24 months
  Compare percent BMD change 12 and 24 months after TKA at the distal femur, 25 percent region of interest between all robotic vs manual implants.

SECONDARY OUTCOMES:
Percent Change in Bone Mineral Density within 15 percent of the region of interest at 12 and 24 months post TKA: All Participants | 12 months, 24 months
  Secondary endpoint is to estimate percent BMD change 12 and 24 months after TKA at the distal femur and the proximal tibia, 15 percent region of interest, reported for all participants together.
Percent Change in Bone Mineral Density within 15 percent of the region of interest at 12 and 24 months post TKA: Cemented vs Uncemented | 12 months, 24 months
  Compare percent BMD change 12 and 24 months after TKA at the distal femur and the proximal tibia, 15 percent region of interest, reported for cemented vs uncemented implants.
Percent Change in Bone Mineral Density within 15 percent of the region of interest at 12 and 24 months post TKA: Robotic vs Manual | 12 months, 24 months
  Compare percent BMD change 12 and 24 months after TKA at the distal femur and the proximal tibia, 15 percent region of interest, reported for robotic vs manual implants.

OTHER OUTCOMES:
Visual Analog Scale (VAS) for Patient Reported Pain | 2 weeks, 3 months, 12 months, 24 months
  Participants will report pain from 0 (no pain) to 10 (worst possible pain)
Patient Reported Function measured by the Oxford Knee Score (OKS) | 2 weeks, 3 months, 12 months, 24 months
  OKS is a 12-item survey scored from 0-4 for a total possible range of scores from 0-48 where higher scores indicate better function.
Patient Reported Function measured by the Koos Jr Knee Survey | 2 weeks, 3 months, 12 months, 24 months
  A 7-item survey scored from 0-4 with cumulative scores converted to 0-100, where higher scores indicate better knee health.
Patient Reported Function measured by the Forgotten Joint Survey | 2 weeks, 3 months, 12 months, 24 months
  A 12-item survey scored from 0-4 with cumulative scores converted to 0-100, where higher scores indicate better outcomes.
Change in Leg Lean Mass measured by Dual energy x-ray absorptiometry (DXA) | 2 weeks, 3 months, 12 months, 24 months
Change in Leg Lean Mass measured by Bioelectrical impedance spectroscopy (BIS) | 2 weeks, 3 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Nickel, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No